CLINICAL TRIAL: NCT00658723
Title: A Prospective, Randomized, Controlled, Superiority Evaluation of Fibrin Patch as an Adjunct to Control Soft Tissue Bleeding During Abdominal, Retroperitoneal, Pelvic, and Thoracic Surgery
Brief Title: The Fibrin Patch Soft Tissue Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ethicon, Inc. (Industry)
Collaborators: OMRIX Biopharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 400-07-002
Record Dates: First submitted 2008-04-11; First posted 2008-04-15 (Estimated); Results first posted 2014-09-11 (Estimated); Last update posted 2014-09-11 (Estimated); Status verified 2014-09

CONDITIONS: Hemostasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: Fibrin Pad
- 2 (Active Comparator): SURGICEL™ Absorbable Hemostat
  Interventions: Device: SURGICEL™

INTERVENTIONS:
Drug: Fibrin Pad — Fibrin Patch is a sterile bio-absorbable combination product consisting of two constituent parts- a flexible matrix and a coating of two biological components (Human Fibrinogen and Human Thrombin).
  Arms: 1
Device: SURGICEL™ — Absorbable hemostat
  Arms: 2

SUMMARY:
The effectiveness objective of this study is to evaluate whether Fibrin Patch is superior to SURGICEL™ as an adjunct to achieving hemostasis during surgical procedures involving soft tissue bleeding in abdominal, pelvic, retroperitoneal and (non-cardiac) thoracic surgery.

ELIGIBILITY:
Inclusion Criteria:

* Subjects >= 18 years of age, requiring non-emergent, open, abdominal, retroperitoneal, pelvic or thoracic (non-cardiac) surgical procedures
* Presence of an appropriate soft tissue Target Bleeding Site (TBS) as identified intraoperatively by the surgeon
* Subjects must be willing to participate in the study, and provide written informed consent

Exclusion Criteria:

* Subjects with any intra-operative findings identified by the surgeon that may preclude conduct of the study procedure
* Subject with TBS within an actively infected field
* Bleeding site is in, around, or in proximity to foramina in bone, or areas of bony confine
* Subjects with known intolerance to blood products or to one of the components of the study product
* Subjects unwilling to receive blood products
* Subjects with immunodeficiency diseases (including known HIV)
* Subjects who are known, current alcohol and / or drug abusers
* Subjects who have participated in another investigational drug or device research study within 30 days of enrollment
* Female subjects who are pregnant or nursing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 141 (Actual)
Dates: Start 2008-03; Primary Completion 2009-04 (Actual); Study Completion 2009-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James Hart, M.D., Study Director — Ethicon, Inc.
Locations (11):
- United States (11):
  - University of Alabama, Birmingham, Alabama
  - Jacksonville Center for Clinical Research, Jacksonville, Florida
  - Baptist Hosptial, Miami, Florida
  - Emory University Hospital, Atlanta, Georgia
  - Medical College of Georgia, Augusta, Georgia
  - University of Maryland Medical Center, Baltimore, Maryland
  - St. Agnes Healthcare, Inc., Baltimore, Maryland
  - Long Island Jewish Medical Center, New Hyde Park, New York
  - Lehigh Valley Hospital, Allentown, Pennsylvania
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - Weill Medical Colleges of Cornell University - Methodist Hospital, Houston, Texas

REFERENCES:
- [Result] Fischer CP, Bochicchio G, Shen J, Patel B, Batiller J, Hart JC. A prospective, randomized, controlled trial of the efficacy and safety of fibrin pad as an adjunct to control soft tissue bleeding during abdominal, retroperitoneal, pelvic, and thoracic surgery. J Am Coll Surg. 2013 Sep;217(3):385-93. doi: 10.1016/j.jamcollsurg.2013.02.036. PMID 23969113
- [Derived] Corral M, Ferko N, Hollmann S, Hogan A, Jamous N, Batiller J, Shen J. Clinician reported ease of use for a novel fibrin sealant patch for hemostasis: results from four randomized controlled trials. Curr Med Res Opin. 2016;32(2):367-75. doi: 10.1185/03007995.2015.1128405. Epub 2015 Dec 21. PMID 26636489

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 11 clinical centers in the US partipcated in the trial enrolled 141 subjects. The first subject randomized: March 26, 2008 and the last subject completed: April 24, 2009
Pre-assignment Details: The efficacy results are based on the intent-to-treat (ITT) set, which is based on 90 randomized subjects from the two randomized arms - Fibrin Pad Randomized and SURGICEL(TM) Randomized. The Fibrin Pad Non-randomized arm was used for the safety analysis set.
Groups:
- Fibrin Pad Randomized: Fibrin Pad: Fibrin Patch is a sterile bio-absorbable combination product consisting of two constituent parts- a flexible matrix and a coating of two biological components (Human Fibrinogen and Human Thrombin). - Randomized
- SURGICEL™ Randomized: SURGICEL™ Absorbable Hemostat
  SURGICEL™: Absorbable hemostat
- Fibrin Pad Non-randomized: Fibrin Pad: Fibrin Patch is a sterile bio-absorbable combination product consisting of two constituent parts- a flexible matrix and a coating of two biological components (Human Fibrinogen and Human Thrombin). (Non - Randomized)
Period: Overall Study
Arm/Group | Fibrin Pad Randomized | SURGICEL™ Randomized | Fibrin Pad Non-randomized
Started | 60 | 30 | 51
Completed | 56 | 26 | 44
Not Completed | 4 | 4 | 7
Not completed — Lost to Follow-up | 0 | 2 | 2
Not completed — Death | 2 | 1 | 4
Not completed — Scheduling Issue | 1 | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Fibrin Pad All: Fibrin Pad: Fibrin Patch is a sterile bio-absorbable combination product consisting of two constituent parts- a flexible matrix and a coating of two biological components (Human Fibrinogen and Human Thrombin). - Randomized & Non Randomized
- SURGICEL™ Randomized: SURGICEL™ Absorbable Hemostat
- Total: Total of all reporting groups
Arm/Group | Fibrin Pad All | SURGICEL™ Randomized | Total
Number analyzed (Participants) | 111 | 30 | 141
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 63 | 21 | 84
  >=65 years | 48 | 9 | 57
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42 | 10 | 52
  Male | 69 | 20 | 89
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 21 | 5 | 26
  White | 90 | 23 | 113
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 111 | 30 | 141

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Subjects Achieving Hemostatic Success
Description: Proportion of success in achieving hemostasis at 4 minutes after randomization with no re-bleeding requiring treatment during a subsequent 6-minute observation period.
Time Frame: Intra-operative
Measure: Number; unit: percentage of success
Groups:
- Fibrin Pad - Randomized: Fibrin Pad: Fibrin Patch is a sterile bio-absorbable combination product consisting of two constituent parts- a flexible matrix and a coating of two biological components (Human Fibrinogen and Human Thrombin). - Randomized
- SURGICEL: SURGICEL™ Absorbable Hemostat
- Fibrin Pad - Non-Randomized: Fibrin Pad: Fibrin Patch is a sterile bio-absorbable combination product consisting of two constituent parts- a flexible matrix and a coating of two biological components (Human Fibrinogen and Human Thrombin). - Non-Randomized
Arm/Group | Fibrin Pad - Randomized | SURGICEL | Fibrin Pad - Non-Randomized
Number analyzed (Participants) | 60 | 30 | 51
percentage of success | 98.3 | 53.3 | 98.0

2. Secondary Outcome: Proportion of Subjects Achieving Hemostatic Success
Description: The proportion of subjects achieving hemostatic success at 10 minutes following randomization
Time Frame: 10 minutes
Measure: Number; unit: percentage of success
Arm/Group | Fibrin Pad - Randomized | SURGICEL | Fibrin Pad - Non-randomized
Number analyzed (Participants) | 60 | 30 | 51
percentage of success | 98.3 | 73.3 | 100.0

3. Secondary Outcome: Incidence of Treatment Failures
Description: If hemostasis was not achieved within 4 minutes or if bleeding required additional intervention during the 6 minute observation period, the treatment was considered to be a failure.
Time Frame: Intra-operative
Measure: Number; unit: percentage of treatment failure
Arm/Group | Fibrin Pad - Randomized | SURGICEL | Fibrin Pad - Non-randomized
Number analyzed (Participants) | 60 | 30 | 51
percentage of treatment failure | 1.7 | 46.7 | 2.0

4. Secondary Outcome: Incidence of Adverse Events That Are Potentially Related to Bleeding
Description: The types of events that were potentially related to bleeding included operative hemorrhage and re-bleeding of the target bleeding site (TBS).
Time Frame: Intra-operative up to 1 month (+14 days)
Measure: Number; unit: percentage of particpants
Arm/Group | Fibrin Pad - Randomized | SURGICEL | Fibrin Pad - Non-randomized
Number analyzed (Participants) | 60 | 30 | 51
percentage of particpants | 0 | 10 | 0

5. Secondary Outcome: Incidence of Adverse Events That Are Potentially Related to Thrombotic Events
Description: The types of events that were potentially related to thrombotic events included deep vein thrombosis and pulmonary embolism
Time Frame: Intra-operative up to 1 month (+14 days)
Measure: Number; unit: percentage of participants
Arm/Group | Fibrin Pad - Randomized | SURGICEL | Fibrin Pad - Non-randomized
Number analyzed (Participants) | 60 | 30 | 51
percentage of participants | 1.7 | 6.7 | 13.7

6. Secondary Outcome: Incidence of Adverse Events Potentially Related to Transfusion Exposure
Description: The types of events that were potentially related to transfusion exposure could have include hypocalcemia.
Time Frame: Intra-operative up to 1 month (+14 days)
Measure: Number; unit: percentage of particpants
Arm/Group | Fibrin Pad - Randomized | SURGICEL | Fibrin Pad - Non-randomized
Number analyzed (Participants) | 60 | 30 | 51
percentage of particpants | 0 | 0 | 0

7. Secondary Outcome: Incidence of Re-treatment
Description: The outcome measure assess if re-treatment was done after release of manual compression at 4-minutes for subjects not achieving hemostatic success or if re-treatment was done during the 6-minute observation period.
  In the SURGICEL group, 18 subjects had initial hemostatic success at 4 minutes, but 2 of the 18 subjects were re-treated for re-bleeding. In the SURGICEL group, 12 subjects were not hemostatic at 4-minutes and had a re-treatment.
Time Frame: Intra-operative
Measure: Number; unit: participants
Arm/Group | Fibrin Pad - Randomized | SURGICEL | Fibrin Pad - Non-randomized
Number analyzed (Participants) | 60 | 30 | 51
participants
  Total Incidence of Re-treatment | 1 | 14 | 1
  No hemostasis at 4-minutes and re-treated | 1 | 12 | 1
  Achieved hemostasis at 4-mins and re-treated | 0 | 2 | 0

8. Secondary Outcome: Incidence of Adverse Events
Time Frame: 30 days (+14 days)
Measure: Number; unit: % if participants with atleast one AE
Arm/Group | Fibrin Pad All | SURGICEL™ Randomized
Number analyzed (Participants) | 111 | 30
% if participants with atleast one AE | 94.6 | 90.0

ADVERSE EVENTS:
Time Frame: 30-Days (+14 Days)
Description: Adverse Events were collected starting at randomization until 30 day follow-up visit (30-Days (+ 14 days))
Arm/Group | Fibrin Pad All | SURGICEL™ Randomized
Serious Adverse Events (participants affected / at risk) | 40/111 | 15/30
Other Adverse Events (participants affected / at risk) | 105/111 | 27/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Fibrin Pad All (N=111) | SURGICEL™ Randomized (N=30)
ANAEMIA (Blood and lymphatic system disorders) | 1 | 0
LEUKOCYTOSIS (Blood and lymphatic system disorders) | 0 | 1
ACUTE MYOCARDIAL INFARCTION (Cardiac disorders) | 0 | 1
ATRIAL FIBRILLATION (Cardiac disorders) | 0 | 1
CARDIAC ARREST (Cardiac disorders) | 0 | 1
CARDIO-RESPIRATORY ARREST (Cardiac disorders) | 2 | 0
MYOCARDIAL INFARCTION (Cardiac disorders) | 1 | 0
VENTRICULAR TACHYCARDIA (Cardiac disorders) | 1 | 0
GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 1 | 1
GASTROINTESTINAL HYPOMOTILITY (Gastrointestinal disorders) | 1 | 0
ILEUS (Gastrointestinal disorders) | 2 | 0
IMPAIRED GASTRIC EMPTYING (Gastrointestinal disorders) | 0 | 1
INTESTINAL INFARCTION (Gastrointestinal disorders) | 1 | 0
INTESTINAL PERFORATION (Gastrointestinal disorders) | 1 | 0
LOCALISED INTRAABDOMINAL FLUID COLLECTION (Gastrointestinal disorders) | 1 | 0
NAUSEA (Gastrointestinal disorders) | 2 | 0
OESOPHAGEAL PERFORATION (Gastrointestinal disorders) | 1 | 0
PANCREATIC FISTULA (Gastrointestinal disorders) | 0 | 1
RETROPERITONEAL HAEMORRHAGE (Gastrointestinal disorders) | 1 | 0
SMALL INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 3 | 0
VOMITING (Gastrointestinal disorders) | 1 | 0
PYREXIA (General disorders) | 0 | 1
ANAPHYLACTIC REACTION (Immune system disorders) | 1 | 0
ABDOMINAL ABSCESS (Infections and infestations) | 3 | 1
ABSCESS (Infections and infestations) | 1 | 0
BRONCHITIS (Infections and infestations) | 1 | 0
EMPYEMA (Infections and infestations) | 1 | 0
LIVER ABSCESS (Infections and infestations) | 1 | 0
PNEUMONIA (Infections and infestations) | 3 | 0
WOUND INFECTION (Infections and infestations) | 3 | 1
ABDOMINAL WOUND DEHISCENCE (Injury, poisoning and procedural complications) | 0 | 1
GASTROINTESTINAL STOMA COMPLICATION (Injury, poisoning and procedural complications) | 2 | 0
OPERATIVE HAEMORRHAGE (Injury, poisoning and procedural complications) | 1 | 0
PERIPANCREATIC FLUID COLLECTION (Injury, poisoning and procedural complications) | 1 | 0
POSTOPERATIVE ILEUS (Injury, poisoning and procedural complications) | 2 | 3
BODY TEMPERATURE INCREASED (Investigations) | 1 | 0
DEHYDRATION (Metabolism and nutrition disorders) | 5 | 0
FAILURE TO THRIVE (Metabolism and nutrition disorders) | 1 | 0
BACK PAIN (Musculoskeletal and connective tissue disorders) | 1 | 0
FISTULA (Musculoskeletal and connective tissue disorders) | 0 | 1
MALIGNANT NEOPLASM PROGRESSION (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 1 | 0
ALCOHOL WITHDRAWAL SYNDROME (Psychiatric disorders) | 1 | 0
HYDRONEPHROSIS (Renal and urinary disorders) | 1 | 0
RENAL FAILURE ACUTE (Renal and urinary disorders) | 1 | 0
URINARY RETENTION (Renal and urinary disorders) | 2 | 0
ACUTE RESPIRATORY DISTRESS SYNDROME (Respiratory, thoracic and mediastinal disorders) | 1 | 0
ATELECTASIS (Respiratory, thoracic and mediastinal disorders) | 1 | 0
BRONCHOPLEURAL FISTULA (Respiratory, thoracic and mediastinal disorders) | 1 | 2
HYPOXIA (Respiratory, thoracic and mediastinal disorders) | 2 | 0
PNEUMOTHORAX (Respiratory, thoracic and mediastinal disorders) | 1 | 0
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 5 | 1
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 2 | 1
SUBCUTANEOUS EMPHYSEMA (Skin and subcutaneous tissue disorders) | 1 | 0
DEEP VEIN THROMBOSIS (Vascular disorders) | 1 | 0
EMBOLISM (Vascular disorders) | 1 | 0
HYPOTENSION (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Fibrin Pad All (N=111) | SURGICEL™ Randomized (N=30)
ANAEMIA (Blood and lymphatic system disorders) | 19 | 7
LEUKOCYTOSIS (Blood and lymphatic system disorders) | 13 | 5
ATRIAL FIBRILLATION (Cardiac disorders) | 10 | 4
ATRIAL FIBRILLATION (Cardiac disorders) | 4 | 2
TACHYCARDIA (Cardiac disorders) | 16 | 4
CONSTIPATION (Gastrointestinal disorders) | 13 | 4
DIARRHOEA (Gastrointestinal disorders) | 7 | 1
DYSPEPSIA (Gastrointestinal disorders) | 3 | 2
ILEUS (Gastrointestinal disorders) | 11 | 4
NAUSEA (Gastrointestinal disorders) | 46 | 14
VOMITING (Gastrointestinal disorders) | 11 | 2
CHEST PAIN (General disorders) | 2 | 2
OEDEMA (General disorders) | 1 | 3
PAIN (General disorders) | 18 | 5
PYREXIA (General disorders) | 22 | 12
ABDOMINAL ABSCESS (Infections and infestations) | 3 | 2
ABDOMINAL INFECTION (Infections and infestations) | 1 | 3
PNEUMONIA (Infections and infestations) | 8 | 3
URINARY TRACT INFECTION (Infections and infestations) | 7 | 1
WOUND INFECTION (Infections and infestations) | 5 | 1
OPERATIVE HAEMORRHAGE (Injury, poisoning and procedural complications) | 1 | 3
POSTOPERATIVE ILEUS (Injury, poisoning and procedural complications) | 2 | 3
PROCEDURAL HYPOTENSION (Injury, poisoning and procedural complications) | 4 | 3
URINE OUTPUT DECREASED (Investigations) | 6 | 0
DEHYDRATION (Metabolism and nutrition disorders) | 5 | 0
FLUID OVERLOAD (Metabolism and nutrition disorders) | 7 | 3
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 26 | 6
HYPOCALCAEMIA (Metabolism and nutrition disorders) | 13 | 8
HYPOGLYCAEMIA (Metabolism and nutrition disorders) | 1 | 2
HYPOKALAEMIA (Metabolism and nutrition disorders) | 29 | 8
HYPOMAGNESAEMIA (Metabolism and nutrition disorders) | 44 | 15
HYPONATRAEMIA (Metabolism and nutrition disorders) | 6 | 1
HYPOPHOSPHATAEMIA (Metabolism and nutrition disorders) | 24 | 15
HYPOVOLAEMIA (Metabolism and nutrition disorders) | 9 | 0
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 1 | 2
ANXIETY (Psychiatric disorders) | 5 | 2
CONFUSIONAL STATE (Psychiatric disorders) | 5 | 0
INSOMNIA (Psychiatric disorders) | 8 | 5
ATELECTASIS (Respiratory, thoracic and mediastinal disorders) | 20 | 6
BRONCHOPLEURAL FISTULA (Respiratory, thoracic and mediastinal disorders) | 6 | 2
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 5 | 2
HYPOXIA (Respiratory, thoracic and mediastinal disorders) | 5 | 2
PHARYNGOLARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 5 | 1
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 17 | 5
PNEUMOTHORAX (Respiratory, thoracic and mediastinal disorders) | 13 | 2
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 5 | 1
PULMONARY OEDEMA (Social circumstances) | 6 | 1
RHONCHI (Respiratory, thoracic and mediastinal disorders) | 6 | 4
PRURITUS (Skin and subcutaneous tissue disorders) | 14 | 3
SUBCUTANEOUS EMPHYSEMA (Skin and subcutaneous tissue disorders) | 5 | 2
HYPERTENSION (Vascular disorders) | 13 | 2
HYPOTENSION (Vascular disorders) | 13 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days